CLINICAL TRIAL: NCT02647099
Title: A Randomized Double-blind Placebo-controlled Study With ASA Treatment in Colorectal Cancer Patients With Mutations in the PI3K Signaling Pathway
Brief Title: Adjuvant Low Dose Aspirin in Colorectal Cancer
Acronym: ALASCCA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Anna Martling (Other)
Collaborators: Uppsala University Hospital (Other); Skane University Hospital (Other)
Responsible Party: Sponsor-Investigator, Anna Martling, Professor, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 921-2014-7074
Record Dates: First submitted 2016-01-05; First posted 2016-01-06 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Colorectal Cancer
Keywords: Aspirin; PI3K signaling pathway
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aspirin (Active Comparator): One tablet acetylsalicylic acid (ASA) 160 mg, orally once daily for three years
  Interventions: Drug: Acetylsalicylic acid
- Placebo (Placebo Comparator): One tablet placebo orally once daily for three years
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetylsalicylic acid
  Other Names: ASA, aspirin
  Arms: Aspirin
Drug: Placebo
  Arms: Placebo

SUMMARY:
ALASCCA is a randomized, parallel group, double blind, multicenter, placebo-controlled, biomarker-based study of adjuvant treatment with low dose aspirin in patients with colorectal cancer. Hypothesis is that patients diagnosed with colorectal cancer and somatic mutations in PI3K pathway can significantly improve survival if treated with low dose aspirin.

DETAILED DESCRIPTION:
Patients with colorectal cancer clinical stage I-III will be screened for inclusion at the time of tumor surgery (at time of routine patient visit before elective surgery or postoperatively within 12 weeks in case of emergency procedure or if screening was missed preoperatively). After inclusion and when surgery is performed, patients with PIK3 mutations and stage II and III tumors will be randomized to receive 160 mg aspirin or placebo orally.

Last date for randomization and start of treatment is 12 weeks postoperatively. The treatment can be administered alone or in combination with adjuvant chemotherapy. The choice of any adjuvant chemotherapy is made by the Investigator and should follow the guidelines in the National Care Program. The treatment will be administered for 3 years. There will be a follow-up period for two years. Outside the trial, the patient will be treated according to standard care at the site.

A phone contact will be made 3 months after the randomization visit and thereafter every 6th month. The patients will also visit the site 6 months after randomization and thereafter every 6th month i.e. the patients will be in contact with the site every 3rd month. There will also be a visit/phone contact at the end of the follow-up period.

The primary objective is to determine whether adjuvant treatment with 160mg ASA once daily for 3 years can improve time to recurrence in participants with colorectal cancer with somatic alternations in the PI3K singling pathway.

UPDATE: New dimensional analysis and power calculation, 19th October 2020:

A total of 3900 patients will be screened in order to include 300 patients with PIK3CA (Exon 9 and 20) mutated tumors in each treatment arm (Group A). With an estimated 10 % drop-out rate, 150 patients will be randomized in each arm. This also includes approximately 15 % of the patients that will be excluded due to tumor stage 1.

An additional 300 patients with mutations in other PI3K pathway genes PIK3CA (other than exon 9 and 20), PIK3R1 or PTEN will also be randomized in each arm and will be treated as a separate group in the analyses (Group B). With an estimated 10 % drop-out rate, 150 patients will be randomized in each arm.

Patients already treated with ASA at inclusion will be included in an observation group.

An interim analysis will be made on safety i.e incidence and type of serious bleeding complication grade > 1 after 12 months. An independent safety data monitoring committee will be responsible for evaluating and follow-up of the safety.

ELIGIBILITY:
Inclusion Criteria:

* Tumor with somatic alterations in PIK3CA, PIK3R1 or PTEN
* Colon or rectal cancer tumor stage II-III
* Radical surgery according to surgeon and pathologist
* Karnofsky performance status ≥60%
* Platelets ≥ 100 x 109 / L
* Clean Colonoscopy or Computed Tomography (CT) colon within 3 months preoperatively or postoperatively but before randomization
* Patient able to swallow tablets
* Patient able to understand and sign written informed consent

Exclusion Criteria:

* Hereditary colorectal cancer linked to familial colonic polyposis or Lynch syndrome
* Inflammatory bowel disease (Crohn's disease or ulcerative colitis)
* Distant metastases
* Other cancers (excluding colorectal cancer or other skin cancer than melanoma) within 3 years from screening
* Known bleeding diathesis (such as hemophilia)
* Concomitant antiplatelet therapy (eg clopidrogrel or ticlopidine) or anticoagulant therapy (warfarin or low molecular weight heparin). Post-operative treatment with low molecular weight heparin must be withdrawn before administration of study treatment
* Active gastritis or peptic ulcer, or significant surgical post-op bleeding, within the previous three months assessed at screening and randomization
* Ongoing regular use of corticosteroids, Nonsteroidal Anti-Inflammatory Drug (NSAID)
* Uncontrolled hypertension according to Investigator's judgment
* Clinically significant liver impairment according to Investigators judgment
* Existing renal failure according to Investigator's judgment. Renal failure with decreased creatinine clearance <60 should lead to consultation with a nephrologist.
* Significant medical illness that would interfere with study participation
* Pregnancy or breastfeeding females
* Known allergy to NSAIDs or ASA
* Current participation in another clinical trial that will be in conflict with the present study
* Patients who are unlikely to comply with the protocol (e.g. uncooperative attitude, inability to return for subsequent visits) and/or otherwise considered by the Investigator to be unlikely to complete the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2016-04-07 (Actual); Primary Completion 2024-08 (Actual); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Time To Recurrence (TTR) | 3 years
  Defined as local recurrence, distant metastases or death from same cancer.

SECONDARY OUTCOMES:
Disease free survival (DFS) | 3 years
Overall survival (OS) | 3 years
Frequency and severity of adverse events (AE) | 1 year and 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Anna Martling, Professor, Principal Investigator — Karolinska Institutet
Locations (32):
- Denmark (3):
  - Aarhus University Hospital, Aarhus
  - Randers Regional Hospital, Randers
  - Viborg Region Hospital, Viborg
- Finland (2):
  - Jorvi Hospital, Espoo
  - Meilahti Tower Hospital, Helsinki
- Norway (4):
  - Akershus University Hospital, Oslo
  - Stavanger University Hospital, Stavanger
  - University Hospital of North Norway, Tromsø
  - St Olavs Hospital, Trondheim
- Sweden (23):
  - Falu Hospital, Falun
  - Eastern Hospital, Gothenburg
  - Ryhov Hospital, Jönköping
  - Blekinge Hospital (Karlskrona-Karlshamn), Karlskrona
  - Karlstad Central Hospital, Karlstad
  - Linköping University Hospital, Linköping
  - Sunderby Hospital, Luleå
  - Skåne University Hospital, Malmo
  - Mora Hospital, Mora
  - Vrinnevi Hospital, Norrköping
  - Örebro University Hospital, Örebro
  - Skaraborg Hospital, Skövde
  - Capio S:t Göran Hospital, Stockholm
  - Danderyd Hospital, Stockholm
  - Ersta Hospital, Stockholm
  - Karolinska University Hospital, Stockholm
  - South Hospital, Stockholm
  - Sundsvall Regional Hospital (Sundsvall-Härnösand), Sundsvall
  - Northern Älvsborg County Hospital, Trollhättan
  - University Hospital of Umeå, Umeå
  - Uppsala University Hospital, Uppsala
  - Västerås Central Hospital, Västerås
  - Ystad Hospital, Ystad

REFERENCES:
- [Derived] Martling A, Hed Myrberg I, Nilbert M, Gronberg H, Granath F, Eklund M, Oresland T, Iversen LH, Haapamaki C, Janson M, Westberg K, Segelman J, Ersson U, Prytz M, Angenete E, Bergstrom R, Mayrhofer M, Glimelius B, Lindberg J; ALASCCA Study Group. Low-Dose Aspirin for PI3K-Altered Localized Colorectal Cancer. N Engl J Med. 2025 Sep 18;393(11):1051-1064. doi: 10.1056/NEJMoa2504650. PMID 40961426

DOCUMENTS (2):
  • Study Protocol (2021-01-25): https://cdn.clinicaltrials.gov/large-docs/99/NCT02647099/Prot_001.pdf
  • Statistical Analysis Plan (2024-08-28): https://cdn.clinicaltrials.gov/large-docs/99/NCT02647099/SAP_002.pdf